CLINICAL TRIAL: NCT01881529
Title: A Non-Interventional Pilot Study Assessing Whether Lysyl Oxidase-like 2 (LOXL2) is Present in Subjects With Scleroderma
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-321-0108
Record Dates: First submitted 2013-06-05; First posted 2013-06-19 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Limited Scleroderma; Diffuse Scleroderma
Keywords: limited scleroderma; diffuse scleroderma; Sclerosis; Progressive; Limited
MeSH Terms: conditions — Scleroderma, Limited; Scleroderma, Diffuse; Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * 5 mL blood draw for LOXL2 testing
  * 2 Punch Skin Biopsies (one near the scleroderma lesion, the other from normal skin)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Limited Scleroderma
- Diffuse Scleroderma

SUMMARY:
To treat patients with scleroderma by blocking the expression of LOXL2. The investigators first need to confirm (through observation) that LOXL2 is overexpressed in disease.

DETAILED DESCRIPTION:
Scleroderma is a chronic skin-hardening disease. There are two types of scleroderma. The first type is called limited cutaneous scleroderma, where disrupted blood flow causes skin discoloration and sometimes patients experience high blood pressure in their arteries. The second type is called diffuse cutaneous scleroderma and it is much more aggressive, affecting a larger area of skin causing organ damage. This study will determine if the disease is associated with an elevated expression of LOXL2 levels in tissue samples from patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Documented diagnosis of scleroderma
* Willing and able to provide written informed consent

Exclusion Criteria:

* Use of experimental therapies within 28 days prior to Screening.
* Aspirin use > 81 mg daily within 1 week prior to Screening.
* Any lab abnormality or concurrent medical condition that, in the opinion of the investigator would make the patient ineligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with documented diagnoses of scleroderma will be enrolled into one of two cohorts, depending upon the subject's diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Summarized the number and percentage of subjects with elevated LOXL2 levels | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, MD, Study Director — Gilead Sciences
Locations (1):
- St Vincent's Centre for Applied Medical Research, Darlinghurst, New South Wales, Australia